CLINICAL TRIAL: NCT04140773
Title: The Effect of D-serine as add-on Therapy in Recent-onset Psychosis
Acronym: DROP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor participant recruitment
Sponsor: Dragos Inta (Other)
Responsible Party: Sponsor-Investigator, Dragos Inta, Prof. Dr. med., Psychiatric Hospital of the University of Basel
Organization: Psychiatric Hospital of the University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-01699
Record Dates: First submitted 2019-10-18; First posted 2019-10-28 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Psychotic Disorder
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-serine group (Experimental): Oral administration of 2g D-serine per day, for 6 weeks.
  Interventions: Dietary Supplement: D-serine
- Placebo group (Placebo Comparator): Oral administration of 2g Placebo (Mannitol) per day, for 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: D-serine — Capsule D-serine
  Arms: D-serine group
Other: Placebo — Capsule D-serine
  Arms: Placebo group

SUMMARY:
In psychotic disorders, negative symptoms and cognitive impairment are difficult to treat with antipsychotics, which are mostly effective for positive symptoms. However, it is important that negative symptoms and cognitive impairment are treated as well, as they both play a large part in the acute episode and long-term course of schizophrenia outcome. Previous studies have used D-serine as add-on treatment in patients with psy-chotic disorders and high-risk patients, with positive results. So far, no study has investigated the effects in a sample of recent-onset psychosis patients.

Therefore, this study will include 30 patients (18-50 years old) with recent-onset psychosis. In addition to their regular treatment, patients will receive either D-serine (2 g/d) or placebo for 6 weeks. D-serine is an amino-acid naturally occurring in the brain which is prescription-free available as nutritional supplement.

The primary outcome measure is total score on the Positive and Negative Syndrome Scale (PANSS). Secondary measure-ments include PANSS subscales, neurocognitive tests, (f)MRI, and EEG

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50
* Recent onset psychosis (< 5 years of overt psychotic symptoms)
* Able to read and understand study procedures and participant's information

Exclusion Criteria:

* Clozapine use
* Suicidal ideation
* Psychotic disorders and symptoms associated with general medical conditions or substance abuse
* BMI > 30
* Renal impairment (history and creatin levels (< 80 ug/L for woman and < 97 ug/L for men))
* Hearing impairment
* Current or past (< 6 months) enrolment in another clinical trial with the primary outcome to improve symptoms
* Pregnant or lactating women (pregnancy test)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Total symptom severity | change from baseline to 6 weeks
  total score on the Positive and Negative Syndrome Scale (PANSS). Lower scores indicate better outcome (min. 30 - max. 120).

SECONDARY OUTCOMES:
Subscales symptom severity | change from baseline to 6 weeks
  Subscores (5-factor model) on the Positive and Negative Syndrome Scale (PANSS). Lower scores indicate better outcome.
Symptom severity and treatment response | change from baseline to 6 weeks
  measured with the Clinical Global Impression Scale (CGI), lower scores indicate a better outcome
Resting-state microstates | change from baseline to 6 weeks
  measured with resting-state electroencephalography (EEG). large-scale neural networks are investigated with EEG microstates Ocillations in the theta-band (4-7 Hz) and gamma-band (>30 Hz) will be assessed.
  measured with resting-state electroencephalography (EEG). Ocillations in the theta-band (4-7 Hz) and gamma-band (>30 Hz) will be assessed.
Mismatch Negativity (MMN) | change from baseline to 6 weeks
  measured with EEG
Intelligence | change from baseline to 6 weeks
  Part of neurocognitive testing. Higher scores indicate better outcome.
Attention and processing speed | change from baseline to 6 weeks
  Part of neurocognitive testing. Higher scores indicate better outcome.
Executive functioning | change from baseline to 6 weeks
  Part of neurocognitive testing. Higher scores indicate better outcome.
Memory | change from baseline to 6 weeks
  Part of neurocognitive testing. Higher scores indicate better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- UPK Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No